CLINICAL TRIAL: NCT02328469
Title: Prospective Study of the Etiology, Pathogenesis, Clinical Picture and Outcome of Aseptic Meningitis in Slovenia
Brief Title: Aseptic Meningoencephalitis in Slovenia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Slovenian Research Agency (Other); University of Ljubljana School of Medicine, Slovenia (Other); Harvard University (Other)
Responsible Party: Principal Investigator, Franc Strle, MD PhD, University Medical Centre Ljubljana
Other Study IDs: mgt-0614
Record Dates: First submitted 2014-05-27; First posted 2014-12-31 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Aseptic Meningitis
Keywords: aseptic meningitis; tick-borne encephalitis; Lyme neuroborreliosis; inflammation; outcome
MeSH Terms: conditions — Meningitis, Aseptic; Encephalitis, Tick-Borne; Lyme Neuroborreliosis; Inflammation | interventions — Ceftriaxone; Doxycycline; Surveys and Questionnaires; Acyclovir

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of full blood, serum and plasma will be collected and retained in deep freezer for further analyses.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- unidentified aseptic meningitis: Patients with etiologically unidentified aseptic meningitis will be treated with symptomatic therapy and will be asked to complete a questionnaire.
  Interventions: Drug: symptomatic therapy; Other: questionnaire
- tick-borne encephalitis: Patient with aseptic meningitis in whom serological diagnosis of tick-borne encephalitis will be established. Patients will be treated with symptomatic therapy and will be asked to complete a questionnaire.
  Interventions: Drug: symptomatic therapy; Other: questionnaire
- Lyme neuroborreliosis: Patients with acute aseptic meningitis in whom Lyme neuroborreliosis will be proven or suspected according to microbiological criteria. Patients will be treated with antibiotic therapy (ceftriaxone or doxycycline) and will be asked to complete a questionnaire.
  Interventions: Drug: symptomatic therapy; Drug: Ceftriaxone or Doxycycline; Other: questionnaire
- healthy controls: Patients will be asked to refer a spouse to serve as a control . If unmarried they will be asked to refer a family member or a friend of +/- 5 years to serve as a control.
  Interventions: Drug: symptomatic therapy; Other: questionnaire
- identified aseptic meningitis: Patients with microbiologically identified cause of acute aseptic meningitis/meningoencephalitis will receive symptomatic therapy. If the identified causative agent will be Herpes Simplex Virus or Varicella Zoster Virus, patients will be treated with acyclovir and will be asked to complete a questionnaire.
  Interventions: Drug: symptomatic therapy; Other: questionnaire; Drug: Acyclovir

INTERVENTIONS:
Drug: symptomatic therapy — patients will receive symptomatic therapy with antipyretics, analgetics, antiemetics and parenteral hydration: metamizole, paracetamol, thiethylperazine, saline
Drug: Ceftriaxone or Doxycycline — beside symptomatic therapy (metamizole, paracetamol, thiethylperazine, saline), patients with proven or probable Lyme neuroborreliosis will be treated with ceftriaxone 2 g intravenously once daily for 14 days OR doxycycline 100 mg orally twice daily for 14 days
  Groups: Lyme neuroborreliosis
Other: questionnaire — Control subjects will be asked to answer a questionnaire asking about the presence and frequency of nonspecific symptoms.
Drug: Acyclovir — Patients will be treated with intravenous acyclovir 10 mg per kg three times daily for 14 to 21 days.
  Groups: identified aseptic meningitis

SUMMARY:
The main objective of this study is:

* to establish etiology of acute aseptic meningitis/meningoencephalitis in Slovenia
* to assess the clinical course and outcome of tick-borne encephalitis and Lyme neuroborreliosis
* to characterize the inflammatory proteins, gene polymorphisms, and transcriptome profiles in patients with tick-borne encephalitis and Lyme neuroborreliosis

ELIGIBILITY:
Inclusion Criteria:

* clinical picture compatible with aseptic meningitis/meningoencephalitis
* age 18 years or older
* clear cerebrospinal fluid on macroscopic examination
* cerebrospinal pleocytosis (> 5 x 106 white blood cells per liter)

Exclusion Criteria:

* younger than 18 years
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult patients with acute aseptic meningitis/meningoencephalitis
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2014-06; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Changes in selected clinical parameters in patients with acute aseptic meningitis/meningoencephalitis | at enrollment and during 12 months follow-up
  Selected clinical parameters (presence or absence of headache, nausea, vomiting, neurologic symptoms, maximal temperature, etc) in aseptic meningitis/meningoencephalitis patients at enrollment (at admission to hospital) and at follow-up visits: on day 7 or on day of discharge from hospital, on day 14, at 2, 6, and 12 months.
Changes in selected laboratory parameters in patients with acute aseptic meningitis/meningoencephalitis | at enrollment and during 12 months follow-up
  Selected laboratory parameters (complete blood count, biochemistry test results) in aseptic meningitis/meningoencephalitis patients at enrollment (at admission to hospital) and at follow-up visits: on day 7 or on day of discharge from hospital, on day 14, at 2, 6, and 12 months.
Changes in selected microbiologic parameters in patients with acute aseptic meningitis/meningoencephalitis | at enrollment and during 12 months follow-up
  Selected microbiologic parameters (anti Borrelia burgdorferi immunoglobulin M and G in serum and cerebrospinal fluid results, polymerase chain reaction for enteroviruses, herpes simplex virus type 1 and 2 in cerebrospinal fluid results) in aseptic meningitis/meningoencephalitis patients at enrollment (at admission to hospital) and anti Borrelia burgdorferi immunoglobulin M and G in serum at follow-up visits: at 2, 6, and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Franc Strle, MD, PhD, Study Chair — UMC Ljubljana; Daša Stupica, MD, PhD, Principal Investigator — UMC Ljubljana
Locations (2):
- Slovenia (2):
  - Department of Infectious Diseases, University Medical Center Ljubljana, Ljubljana, Slovenia, Ljubljana
  - UMC Ljubljana, Department of Infectious Diseases, Ljubljana